CLINICAL TRIAL: NCT06489158
Title: Observation of Exhaled VOC Biomarkers Characteristics in Admitted Women with Breast Ultrasound BI-RADS 4 Grade
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-BCVOC200
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Exhaled samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Benign breast disease: The accuracy of VOCs indicators and ultrasound 4a/4b/4c diagnosis will be compared in determining benign and malignant diseases based on pathological gold standards.
  Interventions: Diagnostic Test: Detect VOCs in exhaled gas
- Breast Cancer: The accuracy of VOCs indicators and ultrasound 4a/4b/4c diagnosis will be compared in determining benign and malignant diseases based on pathological gold standards.
  Interventions: Diagnostic Test: Detect VOCs in exhaled gas

INTERVENTIONS:
Diagnostic Test: Detect VOCs in exhaled gas — The exhaled gas of the patients should be collected within one week before surgery and be tested within 24 hours after enrollment. Then receive treatment according to the existing diagnosis and treatment process.

SUMMARY:
1. Explore VOCs indicators that can effectively distinguish between benign and malignant breast diseases.
2. The accuracy of VOCs indicators and ultrasound 4a/4b/4c diagnosis will be compared in determining benign and malignant diseases based on pathological gold standards.

DETAILED DESCRIPTION:
Inclusion Criteria:

Ultrasound examination within 3 months clearly indicates that breast lesions are BI-RADs4a/4b/4c Surgical treatment within one week after Exhaled VOC test informed consent form should be signed

Exclusion Criteria:

Male Women who have been diagnosed as breast cancer by puncture Individuals with unclear BI-RADs level information by breast ultrasound, including but not limited to BI-RADs 4/3-4a/4a-b/4b-c Pregnant or lactating women A positive smoking history within one year Medical history of malignant tumor, including but not limited to breast cancer (excluding skin basal cell carcinoma) The past history of metabolic diseases, including diabetes, gout, etc Respiratory diseases that have been clearly diagnosed in the past, such as asthma and chronic obstructive pulmonary emphysema, are not suitable for participation in the study Previously diagnosed digestive system diseases, such as Helicobacter pylori positivity and gastric ulcers, are not suitable for participation in the study Combination application of drugs related to the treatment of elderly dementia Possible cases which researchers believe it is not suitable for this clinical research

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound examination within 3 months clearly indicates that breast lesions are BI-RADs4a/4b/4c
* Surgical treatment within one week after Exhaled VOC test
* informed consent form should be signed

Exclusion Criteria:

* Male
* Women who have been diagnosed as breast cancer by puncture
* Individuals with unclear BI-RADs level information by breast ultrasound, including but not limited to BI-RADs 4/3-4a/4a-b/4b-c
* Pregnant or lactating women
* A positive smoking history within one year
* Medical history of malignant tumor, including but not limited to breast cancer (excluding skin basal cell carcinoma)
* The past history of metabolic diseases, including diabetes, gout, etc
* Respiratory diseases that have been clearly diagnosed in the past, such as asthma and chronic obstructive pulmonary emphysema, are not suitable for participation in the study
* Previously diagnosed digestive system diseases, such as Helicobacter pylori positivity and gastric ulcers, are not suitable for participation in the study
* Combination application of drugs related to the treatment of elderly dementia
* Possible cases which researchers believe it is not suitable for this clinical research

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with BI-RADs 4 breast lesions by ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Exhaled VOC Biomarkers | 1 year
  The relationship between exhaled VOC and breast cancer grading will be studied. 168 patients with With Breast Ultrasound BI-RADS 4 Grade were enrolled. Exhale gas was collected and tested using mass spectrometer. Exhaled VOC biomarkers characteristics in admitted women with breast ultrasound BI-RADS 4 grade will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- 41 Damucang Hutong, Xicheng District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No